CLINICAL TRIAL: NCT00795665
Title: Phase II Study of Bevacizumab (Avastin) and BCNU for Treatment of Relapsed, High Grade Gliomas
Brief Title: Bevacizumab and Carmustine in Treating Patients With Relapsed or Progressive High-Grade Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 224865; UCDCC#208 (Other: UC Davis); P30CA093373 (NIH)
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Glioma
Keywords: adult anaplastic astrocytoma; adult glioblastoma; adult gliosarcoma; adult giant cell glioblastoma; adult anaplastic oligodendroglioma; adult mixed glioma; recurrent adult brain tumor
MeSH Terms: conditions — Glioma; Astrocytoma; Glioblastoma; Gliosarcoma; Oligodendroglioma; Brain Neoplasms | interventions — Bevacizumab; Carmustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab and Carmustine (Experimental)
  Interventions: Drug: bevacizumab; Drug: carmustine

INTERVENTIONS:
Drug: bevacizumab — Bevacizumab (10 mg/kg) will be given intravenously every other week starting one week before the first dose of BCNU. Treatment with both BCNU and bevacizumab for 6-months, after which the participant may continue to receive bevacizumab every 2 weeks for a maximum of one year and three additional cycles of BCNU.
  Other Names: Avastin
Drug: carmustine — BCNU (200 mg/m2), will be given over 4 hours as a continuous intravenous infusion every 8 weeks. Treatment with both BCNU and bevacizumab for 6-months, after which the participant may continue to receive bevacizumab every 2 weeks for a maximum of one year and three additional cycles of BCNU.
  Other Names: BCNU

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Drugs used in chemotherapy, such as carmustine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bevacizumab together with carmustine may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving bevacizumab together with carmustine works in treating patients with relapsed or progressive high-grade glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the 6-month progression-free survival of patients with relapsed or progressive high-grade gliomas treated with bevacizumab and carmustine.

Secondary

* To evaluate the radiographic response to this regimen as measured by MRI and PET scan with image fusion.
* To utilize novel brain imaging to differentiate between a radiographic response due to tumor shrinkage and a radiographic response due to decreased vasogenic edema.
* To evaluate the safety and toxicity of this regimen in these patients.
* To evaluate the overall survival of these patients.

OUTLINE: Patients receive bevacizumab IV on days -7, 8, 22, 36, and 50 of course 1 and on days 8, 22, 36, and 50 of all subsequent courses. Patients also receive carmustine IV over 4 hours on day 1. Treatment repeats every 56 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed GBM, anaplastic astrocytoma, anaplastic oligoastrocytoma or anaplastic oligodendroglioma.
* Disease progression (confirmed by MRI, PET or both) after radiation therapy
* At least 28 days have elapsed since chemotherapy, major surgery or radiation therapy.
* No other malignancy within 3 years except for non-melanomatous skin cancer or in situ cervical cancer.
* Karnofsky performance score at least 70
* Platelet count ≥ 130/mm3.
* Absolute neutrophil count ≥ 1500/mm3
* Calculated creatinine clearance greater than 45 mg/dl
* AST < 2 times the upper limit of normal
* Bilirubin < 1.5 times the upper limit of normal
* Ability to give signed informed consent
* Patients must be 18 years of age or older.

Exclusion Criteria:

* Prior intravenous or oral nitrosoureas (BCNU, CCNU) or prior VEGF targeted therapy including bevacizumab. No more than two prior chemotherapy regimens are allowed. Prior or current steroid use is allowed.
* Evidence of CNS hemorrhage
* Requirement for therapeutic anticoagulation
* Any grade 3 or greater hemorrhage within the previous 28 days
* Active inflammatory bowel disease
* Inadequately controlled hypertension
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to study enrollment
* History of stroke or transient ischemic attack within 6 months prior to study enrollment
* Significant vascular disease
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Serious, non-healing wound, ulcer, or bone fracture
* Proteinuria at screening
* Pregnant (or lactating). Use of effective means of contraception in subjects of child-bearing potential
* Prior organ transplantation
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* Known acquired immune deficiency syndrome (AIDS) or HIV positive status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert T. O'Donnell, MD, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Cancer Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bevacizumab and Carmustine
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab and Carmustine
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Time from first day of treatment to the first observation of disease progression or death due to any cause (up to 7 years).
Population: Procedure for fusing PET and MRI images could not be performed; as such the volumetrics of areas of tumor versus cerebral edema could not be analyzed or interpreted, therefore, no data can be reported.
Arm/Group | Bevacizumab and Carmustine
Number analyzed (Participants) | 0

2. Secondary Outcome: Radiographic Response to Therapy
Description: Response measured using MRI and PET with image fusion
Time Frame: One year
Population: as for outcome 1
Arm/Group | Bevacizumab and Carmustine
Number analyzed (Participants) | 0

3. Secondary Outcome: Differentiate a Radiographic Response Due to Tumor Shrinkage From a Radiographic Response Due to Decreased Vasogenic Edema
Description: Measurements made by novel brain imaging
Time Frame: One year
Population: as for outcome 1
Arm/Group | Bevacizumab and Carmustine
Number analyzed (Participants) | 0

4. Secondary Outcome: Safety and Toxicity
Description: Subjects will be assessed clinically for toxicity prior to, during, and after each infusion. NCI CTCAE 3.0 Common Terminology Criteria (CTC) for Adverse Events for toxicity and Adverse Event Reporting will be utilized.
Time Frame: One year
Population: as for outcome 1
Arm/Group | Bevacizumab and Carmustine
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Time Frame: Time from first day of treatment to time of death due to any cause (up to 7 years).
Population: as for outcome 1
Arm/Group | Bevacizumab and Carmustine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 36 months.
Arm/Group | Bevacizumab and Carmustine
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab and Carmustine (N=7)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 3
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 2
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 2
Cystitis (Renal and urinary disorders) | 2
Edema limbs (Blood and lymphatic system disorders) | 2
Fatigue (General disorders) | 3
Flu-like syndrome (General disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 4
Hemoglobin decreased (Blood and lymphatic system disorders) | 1
Hemorrhage - subconjunctival (Blood and lymphatic system disorders) | 1
Hemorrhage nasal (Blood and lymphatic system disorders) | 1
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Hypertension (Cardiac disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Infection - Other (Ear Abscess) (Metabolism and nutrition disorders) | 1
Infection - Other (Urinary Tract, NOS) (Metabolism and nutrition disorders) | 1
Ischemia cerebrovascular (Nervous system disorders) | 1
Joint pain (Musculoskeletal and connective tissue disorders) | 1
Leukocytes (Blood and lymphatic system disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 4
Nausea (Gastrointestinal disorders) | 1
Neutrophils (Blood and lymphatic system disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (arm) (Musculoskeletal and connective tissue disorders) | 1
Platelet count decreased (Blood and lymphatic system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 5
Pneumonia (Infections and infestations) | 1
Proteinuria (Metabolism and nutrition disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1
Urinary tract infection (Infections and infestations) | 2

LIMITATIONS AND CAVEATS:
The PI has indicated that data were uninterpretable for the outcome measures in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes